CLINICAL TRIAL: NCT02325895
Title: Effect of Dried Plum on Bone and Bone Biomarkers in Older Women
Brief Title: Dried Plums for Bone Health in Older Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Florida State University (Other)
Responsible Party: Principal Investigator, Dr. Shirin Hooshmand, Assistant Professor, San Diego State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 57114A
Record Dates: First submitted 2014-12-11; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Bone Diseases, Metabolic
Keywords: Osteoporosis; Dried plum; functional food
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (0 g Dried plum/day) (No Intervention): Participants only received 400IU of vitamin D and 500mg of calcium daily for 6 months.
- 50 g Dried plum/day (Experimental): Participants received 400IU of vitamin D and 500mg of calcium and 50g of dried plum daily for 6 months.
  Interventions: Other: Dried Plum
- 100 g Dried plum/day (Experimental): Participants received 400IU of vitamin D and 500mg of calcium and 100g of dried plum daily for 6 months.
  Interventions: Other: Dried Plum

INTERVENTIONS:
Other: Dried Plum — Three doses of dried plum (0 g, 50 g and 100g) were used as intervention.
  Arms: 100 g Dried plum/day; 50 g Dried plum/day

SUMMARY:
The objective of the investigators current study was to examine whether 50 g dried plum would be as effective as 100 g dried plum in reversing bone loss in osteopenic older postmenopausal women.

DETAILED DESCRIPTION:
Forty-five randomly assigned into one of three treatment groups: 1) 50g dried plum; 2) 100g dried plum; and 3) control (0g dried plum). All groups received 500mg calcium and 400 IU vitamin D as a daily supplement. Blood samples were collected at baseline, 3 and 6 months to assess biomarkers of bone turnover. Physical activity recall and 3-day food records were obtained at baseline, 3 and 6 months to examine physical activity and dietary confounders as potential covariates

ELIGIBILITY:
Inclusion Criteria:

* BMD t-score of L1-L4 between -1 to -2.5 standard deviation of the mean
* Age 65 to 79

Exclusion Criteria:

* BMD t-score at any site fell below 2.5 standard deviation of the mean
* Subjects treated with calcitonin, bisphosphonates, raloxifene and/or anabolic agents such as parathyroid hormone and growth hormone, or steroids within three months before the start of the study
* Metabolic bone disease, renal disease, cancer, CVD, diabetes mellitus, respiratory disease, gastrointestinal disease, liver disease or other chronic diseases, heavy smoking (more than twenty cigarettes/day) and current use of any prescription medications known to alter bone and calcium metabolism
* Regularly consumed dried plum or prune juice were not included in the study.

Ages: 65 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 6 months

SECONDARY OUTCOMES:
Changes from baseline in bone specific alkaline phosphatase at 3 months and 6 months | baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hooshmand, PhD, Principal Investigator — San Diego State Univeristy

REFERENCES:
- [Derived] Hooshmand S, Kern M, Metti D, Shamloufard P, Chai SC, Johnson SA, Payton ME, Arjmandi BH. The effect of two doses of dried plum on bone density and bone biomarkers in osteopenic postmenopausal women: a randomized, controlled trial. Osteoporos Int. 2016 Jul;27(7):2271-2279. doi: 10.1007/s00198-016-3524-8. Epub 2016 Feb 22. PMID 26902092